CLINICAL TRIAL: NCT02492750
Title: Phase I/II Double Blind Randomized Trial of Lenalidomide/Dexamethasone/Anakinra vs. Lenalidomide/Dexamethasone/Placebo in Patients With Early Stage Multiple Myeloma and High Plasma Cell Growth Rate
Brief Title: Lenalidomide and Dexamethasone With or Without Anakinra in Treating Patients With Early Stage Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MC138B; NCI-2015-01041 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); RV-CL-MM-PI-004334; MC138B (Other: Mayo Clinic); P30CA015083 (NIH)
Record Dates: First submitted 2015-07-06; First posted 2015-07-09 (Estimated); Results first posted 2020-03-25 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2019-06

CONDITIONS: Indolent Plasma Cell Myeloma; Plasma Cell Myeloma; Smoldering Plasma Cell Myeloma
MeSH Terms: conditions — Multiple Myeloma; Smoldering Multiple Myeloma | interventions — Interleukin 1 Receptor Antagonist Protein; Receptors, Interleukin-6; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; Lenalidomide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (lenalidomide, dexamethasone, anakinra) (Experimental): Patients receive lenalidomide PO on days 1-21 and dexamethasone PO on days 1, 8, 15, and 22. Patients also receive anakinra SC on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity
  Interventions: Biological: Anakinra; Drug: Dexamethasone; Other: Laboratory Biomarker Analysis; Drug: Lenalidomide
- Arm B (lenalidomide, dexamethasone, placebo) (Active Comparator): Patients receive lenalidomide and dexamethasone as in Arm A. Patients also receive placebo SC on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Dexamethasone; Other: Laboratory Biomarker Analysis; Drug: Lenalidomide; Other: Placebo

INTERVENTIONS:
Biological: Anakinra — Given SC
  Other Names: Kinaret; Kineret; rIL-1ra; rIL1RN
  Arms: Arm A (lenalidomide, dexamethasone, anakinra)
Drug: Dexamethasone — Given PO
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Fluorodelta; Fortecortin; Gammacorten; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; Visumetazone
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Lenalidomide — Given PO
  Other Names: CC-5013; CC5013; CDC 501; Revlimid
Other: Placebo — Given SC
  Other Names: placebo therapy; PLCB; sham therapy
  Arms: Arm B (lenalidomide, dexamethasone, placebo)

SUMMARY:
This partially randomized phase I/II trial studies the side effects and best dose of anakinra when given together with lenalidomide and dexamethasone in treating patients with early stage multiple myeloma. Biological therapies, such as lenalidomide and anakinra, may stimulate or suppress the immune system in different ways and stop cancer cells from growing. Drugs used in chemotherapy, such as dexamethasone, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. It is not yet known whether lenalidomide and dexamethasone are more effective with or without anakinra in treating patients with multiple myeloma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD)/maximum allowable dose (MAD) of anakinra that can be combined with lenalidomide and dexamethasone. (Phase I) II. To compare the time to progression of the standard treatment arm (lenalidomide/dexamethasone) to the experimental arm (lenalidomide/dexamethasone + anakinra). (Phase II)

SECONDARY OBJECTIVES:

I. To compare the response rate of the standard treatment arm (lenalidomide/dexamethasone) to the experimental arm (lenalidomide/dexamethasone + anakinra).

II. To compare the toxicity of the standard treatment arm (lenalidomide/dexamethasone) to the experimental arm (lenalidomide/dexamethasone + anakinra).

III. To compare the overall survival of the standard treatment arm (lenalidomide/dexamethasone) to the experimental arm (lenalidomide/dexamethasone + anakinra).

OUTLINE: This is a phase I, dose-escalation study of anakinra followed by a phase II study.

PHASE I: Patients receive lenalidomide orally (PO) on days 1-21 and dexamethasone PO on days 1, 8, 15, and 22. Patients also receive anakinra subcutaneously (SC) on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

PHASE II: Patients are randomized to 1 of 2 treatment arms.

ARM A: Patients receive lenalidomide PO on days 1-21 and dexamethasone PO on days 1, 8, 15, and 22. Patients also receive anakinra SC on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ARM B: Patients receive lenalidomide and dexamethasone as in Arm A. Patients also receive placebo SC on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Absolute neutrophil count (ANC) >= 1700/mm^3
* Platelet count >= 100,000/mm^3
* Hemoglobin >= 8.0 g/dL
* Serum glutamic oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) =< 3 x upper limit of normal (ULN)
* Creatinine clearance >= 30 mL/min (as determined by Cockroft-Gault equation)
* Diagnosis of multiple myeloma according to International Myeloma Working Group criteria and one of the following:

  * Smoldering multiple myeloma (SMM)
  * Indolent multiple myeloma (IMM)
  * Newly diagnosed multiple myeloma (MM)
  * Note: patients with lytic disease and anemia are eligible
* High risk disease defined by all of the following:

  * >= 10% bone marrow plasma cells AND
  * Abnormal serum free light chain (FLC) ratio (< 0.26 or > 1.65) by serum FLC assay AND
  * Monotypic plasma cell S-phase >= 0.3%
* Measurable level of M-protein > 1 g/dL on serum protein electrophoresis or > 200 mg of M-protein on a 24 hour urine protein electrophoresis
* Negative tuberculosis (TB) testing (Quantiferon - TB blood test or skin test) =< 7 days prior to registration
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1 or 2
* Provide signed informed consent
* Negative (serum or urine) pregnancy test done =< 7 days prior to registration, for women of childbearing potential only; NOTE: a second pregnancy test must be performed within 24 hours prior to the start of lenalidomide; the subject may not receive lenalidomide until the study doctor has verified that the results of these pregnancy tests are negative
* Willing to return to enrolling institution for follow-up (during the active monitoring phase of the study)
* Willing and able to comply with the requirements of the Revlimid Risk Evaluation and Mitigation Strategy (REMS) program
* Females of childbearing potential must be willing to adhere to the scheduled pregnancy testing as required by the Revlimid REMS program

Exclusion Criteria:

* Prior treatment with any other agent that may affect M-protein =< 30 days prior to registration
* Acute/chronic infections, open wounds, or any active infection requiring intravenous antibiotic therapy =< 12 weeks prior to registration
* Other active malignancy (=< 3 years) prior to registration; exceptions: basal cell skin cancer or carcinoma-in-situ of the cervix or low-risk prostate cancer after curative therapy
* Any of the following:

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception
* New York Heart Association (NYHA) class 3 or 4 congestive heart failure (CHF) symptoms
* Other concurrent chemotherapy, radiotherapy, or any ancillary therapy considered investigational; NOTE: bisphosphonates are allowed while on protocol treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2019-06-05 (Actual); Study Completion 2019-09-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Lust, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase I - Dose Level 1: Participants receive 25 mg lenalidomide PO on days 1-21; SMM and IMM participants receive 20 mg dexamethasone PO on days 1, 8, 15, and 22; Active MM participants receive 40 mg dexamethasone PO on days 1, 8, 15, and 22. Participants also receive the starting dose of 100 mg anakinra SQ every third day. Participants also receive 325 mg aspirin PO per day with food on days 1-28.
- Phase I - Dose Level 2: Participants receive 25 mg lenalidomide PO on days 1-21; SMM and IMM participants receive 20 mg dexamethasone PO on days 1, 8, 15, and 22; Active MM participants receive 40 mg dexamethasone PO on days 1, 8, 15, and 22. Participants also receive 100 mg anakinra SQ every other day. Participants also receive 325 mg aspirin PO per day with food on days 1-28.
- Phase I - Dose Level 3: Participants receive 25 mg lenalidomide PO on days 1-21; SMM and IMM participants receive 20 mg dexamethasone PO on days 1, 8, 15, and 22; Active MM participants receive 40 mg dexamethasone PO on days 1, 8, 15, and 22. Participants also receive 100 mg anakinra SQ every day on days 1-28. Participants also receive 325 mg aspirin PO per day with food on days 1-28.
Period: Overall Study
Arm/Group | Phase I - Dose Level 1 | Phase I - Dose Level 2 | Phase I - Dose Level 3
Started | 4 | 4 | 6
Completed | 4 | 4 | 6
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I - Dose Level 1 | Phase I - Dose Level 2 | Phase I - Dose Level 3 | Total
Number analyzed (Participants) | 4 | 4 | 6 | 14
Age, Continuous [Median (Full Range); unit: years] | 67 [46 to 86] | 62.5 [49 to 76] | 58.5 [35 to 73] | 60 [35 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 1 | 4
  Male | 2 | 3 | 5 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 4 | 6 | 14
  Unknown or Not Reported | 0 | 0 | 0 | 0
ISS Stage of myeloma at diagnosis [Count of Participants; unit: Participants] — International Staging System (ISS) Stage for Multiple Myeloma:
  I: Serum β2 microglobulin < 3.5 mg/l; Serum albumin ≥ 3.5 g/dl; Standard-risk chromosomal abnormalities (CA); Normal LDH II: Not R-ISS stage I or III III: Serum β2 microglobulin ≥ 5.5 mg/L and either; High-risk CA by FISH OR High LDH Population: Data available are summarized here (i.e. participants with missing data are not included in this analysis).
  Participants
    number analyzed (Participants) | 2 | 1 | 6 | 9
    I | 1 | 0 | 5 | 6
    II | 1 | 1 | 1 | 3
ECOG Performance Score at baseline [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group PS Scale: 0)Fully active, able to carry on all pre-disease performance without restriction; 1)Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work; 2)Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours; 3)Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours; 4)Completely disabled. Cannot carry on any selfcare. Totally confined to bed or chair.
  Participants
    0 | 3 | 2 | 6 | 11
    1 | 1 | 2 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing a Dose-limiting Toxicity (DLT)
Description: Number of participants experiencing a dose-limiting toxicity (DLT) is reported below. Dose-limiting toxicity is graded by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I - Dose Level 1 | Phase I - Dose Level 2 | Phase I - Dose Level 3
Number analyzed (Participants) | 4 | 4 | 6
Participants | 0 | 0 | 0
Statistical Analysis 1: Comparison: Phase I - Dose Level 1 vs Phase I - Dose Level 2 vs Phase I - Dose Level 3; Test type: Other; Maximum Tolerated Dose (MTD) Level = 3 — MTD is defined as the dose level below the lowest dose that induces DLT in at least one-third of patients. A total of 6 patients treated at the MTD will be sufficient to identify common toxicities at the MTD

2. Primary Outcome: Number of Participants Who Experienced at Least One Grade 3+ Adverse Events Deemed at Least Possibly Related to Treatment, Graded According to NCI CTCAE Version 4.0
Description: The number of participants who experienced at least one grade 3+ adverse events deemed at least possibly related to treatment, graded according to NCI CTCAE version 4.0, is reported below.
Time Frame: Up to 41 months
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I - Dose Level 1 | Phase I - Dose Level 2 | Phase I - Dose Level 3
Number analyzed (Participants) | 4 | 4 | 6
Participants | 2 | 3 | 3

3. Primary Outcome: Best Response
Description: The following response terms will be used: stringent Complete Response (sCR), complete response (CR), very good partial response (VGPR), partial response (PR), Minimal Response (MR), stable disease (SD), and progressive disease (PD). The International Myeloma Working Group (IMWG) uniform response criteria (Rajkumar et al, 2011) will be used to assess response to therapy. PR defined as: ≥50% reduction of serum M-protein and reduction in 24-hour urinary M-protein by ≥90% or to <200 mg/24hrs; ≥ 50% reduction in the size of soft tissue plasmacytomas. MR defined as: ≥25% but ≤ 49% reduction of serum M protein and reduction in 24-hour urine M-protein by 50-89% which still exceeds 200mg/24 hours; 25-49% reduction in the size of soft tissue plasmacytoma and No increase in the size or number of lytic bone lesions. VGPR defined as: Serum and urine M-protein detectable by immunofixation but not on electrophoresis or ≥90% reduction in serum M-protein and urine M-protein <100 mg/24 h
Time Frame: Up to 41 months
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I - Dose Level 1 | Phase I - Dose Level 2 | Phase I - Dose Level 3
Number analyzed (Participants) | 4 | 4 | 6
Participants
  Partial Response (PR) | 2 | 3 | 3
  Minimal Response (MR) | 1 | 1 | 2
  Very Good Partial Response (VGPR) | 1 | 0 | 1

ADVERSE EVENTS:
Time Frame: Up to 41 months
Arm/Group | Phase I - Dose Level 1 | Phase I - Dose Level 2 | Phase I - Dose Level 3
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4 | 1/6
Serious Adverse Events (participants affected / at risk) | 1/4 | 1/4 | 1/6
Other Adverse Events (participants affected / at risk) | 4/4 | 4/4 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I - Dose Level 1 (N=4) | Phase I - Dose Level 2 (N=4) | Phase I - Dose Level 3 (N=6)
Lung infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I - Dose Level 1 (N=4) | Phase I - Dose Level 2 (N=4) | Phase I - Dose Level 3 (N=6)
Anemia (Blood and lymphatic system disorders) | 4 (60) | 3 (8) | 3 (19)
Constipation (Gastrointestinal disorders) | 2 (23) | 4 (24) | 5 (11)
Diarrhea (Gastrointestinal disorders) | 2 (35) | 3 (12) | 5 (20)
Dry mouth (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (26) | 1 (1) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Fatigue (General disorders) | 4 (71) | 3 (13) | 3 (18)
Injection site reaction (General disorders) | 4 (8) | 4 (12) | 5 (15)
Mucosal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 1 (1) | 0 (0) | 2 (2)
Lymphocyte count decreased (Investigations) | 3 (10) | 3 (13) | 2 (9)
Neutrophil count decreased (Investigations) | 3 (32) | 3 (27) | 5 (24)
Platelet count decreased (Investigations) | 3 (41) | 2 (7) | 0 (0)
White blood cell decreased (Investigations) | 3 (13) | 2 (11) | 2 (16)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (3) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (3)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (5) | 2 (29) | 4 (20)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Delusions (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Euphoria (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 4 (55) | 4 (39) | 5 (28)
Chronic kidney disease (Renal and urinary disorders) | 2 (4) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (6) | 3 (7) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (7) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-19): https://cdn.clinicaltrials.gov/large-docs/50/NCT02492750/Prot_SAP_000.pdf